CLINICAL TRIAL: NCT07202936
Title: Cervical Pre-cancer Treatment Failure Among Women Living With HIV in Zimbabwe: a Cohort Study
Brief Title: Cervical Pre-cancer Treatment Failure Among Women Living With HIV in Zimbabwe
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2023-00923; U01AI069924 (NIH)
Record Dates: First submitted 2025-07-15; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Uterine Cervical Neoplasms; HIV I Infection; HPV Infection
Keywords: Cervical pre-cancer treatment; Women living with HIV; Zimbabwe; DNA methylation
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — * Cervical biopsies within the transformation zone will be obtained from all women as the reference standard.
  * Nurse-collected cervical and self-collected first-void urine samples will be obtained for HPV and DNA methylation testing.
  * Blood will be drawn for CD4 cell count and HIV RNA viral load analyses, and a vaginal swab will be collected for microbiome analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to improve cervical pre-cancer treatment outcomes among women living with HIV (WLWH), particularly in low and middle income countries (LMICs), by generating the evidence needed for post-treatment monitoring guidelines. The main questions it aims to answer are:

* What is the risk of disease recurrence/persistence after cervical pre-cancer treatment among women living with HIV in Zimbabwe?
* What is the predictive value of different human papillomavirus (HPV) and DNA methylation testing strategies for monitoring cervical disease recurrence/persistence after pre-cancer treatment?

Participants will have cervical biopsies taken for histological assessment and cervical samples for HPV genotyping and DNA methylation testing.

Researchers will follow all participating women every six months for 24 months to evaluate post-treatment monitoring and cervical disease outcomes.

DETAILED DESCRIPTION:
Background and Rationale:

Cervical cancer mortality rates in Zimbabwe are among the highest in the world. Cervical cancer disproportionally affects women living with HIV (WLWH). In 2020, the World Health Assembly adopted a strategy to eliminate cervical cancer as a public health problem. To date, global efforts to eliminate cervical cancer have focused on expanding coverage of HPV vaccination, cervical cancer screening, and treatment for cervical pre-cancerous lesions. However, without monitoring treatment outcomes and ensuring that pre-cancerous lesions were successfully removed, the ambitious goal of cervical cancer elimination may not be attainable.

Cervical disease persistence and recurrence after pre-cancer treatment are common in WLWH. Data on the accuracy of post-treatment screening tests to guide clinical management are scarce. In July 2021, the World Health Organization (WHO) released new cervical cancer screening guidelines that propose primary HPV testing for all women. For follow-up of treated WLWH, the WHO guidelines suggest HPV testing at 12 and 24 months and immediate re-treatment for those who test positive. However, HPV is highly prevalent in WLWH, and the predictive value of a positive test for high-risk HPV infection after pre-cancer treatment in WLWH is uncertain but probably low. Therefore, alternative testing strategies such as confirmation of type-specific HPV persistence, extended HPV genotyping, and combining HPV testing with DNA methylation triage need to be explored. DNA methylation occurs as HPV infection progresses to cervical pre-cancer and cancer. Thus, methylation tests may distinguish between transient and persistent HPV infections that will advance to cancer. An advantage of molecular methylation tests is that they can be automated and are less subjective than morphological tests.

Objective(s):

Primary objectives:

* To estimate the risk of persistent/recurrent Cervical Intraepithelial Neoplasia grade 2 or 3 (CIN2+) at 6, 12, 18, and 24 months after pre-cancer treatment.
* To determine the accuracy and predictive value of the following HPV testing strategies in cervical samples for detection of post-treatment CIN2+ recurrence/persistence among WLWH: i) HPV type-specific persistence, ii) HPV genotyping algorithms, iii) DNA methylation testing, and iv) testing for any high-risk HPV.

Main secondary objectives:

* To identify predictors for persistent/recurrent CIN2+.
* To determine the accuracy and predictive value of different HPV and DNA methylation testing strategies in urine samples for detection of post-treatment CIN2+.
* To examine the agreement of HPV and DNA methylation results between cervical and urine samples.

Study design:

The project will analyze data from a prospective cohort study of 250 WLWH aged 18-65 years treated for cervical pre-cancer at the Newlands Clinic Women's Health Centre in Harare, Zimbabwe. The cohort study will follow all women every six months for 24 months to evaluate post-treatment monitoring and cervical disease outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-65 years
* Positive HIV status confirmed through medical records
* Positive test result for any high-risk HPV genotype at preceding cervical cancer screening visit
* Cervical pre-cancer treatment required according to Newlands Clinic guidelines
* Signed informed consent

Exclusion Criteria:

* Women with a history or suspicion of cervical cancer
* Women with a history of total hysterectomy (no cervix)
* Women treated for cervical pre-cancer in the past 12 months
* Pregnant women

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women living with HIV who are high-risk HPV positive and need cervical pre-cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative CIN2+ persistence | 6 months
  Proportion of participants with histologically confirmed CIN2+ at 6 months after pre-cancer treatment
Cumulative CIN2+ persistence | 12 months
  Proportion of participants with histologically confirmed CIN2+ up to 12 months after pre-cancer treatment
Cumulative CIN2+ persistence | 18 months
  Proportion of participants with histologically confirmed CIN2+ up to 18 months after pre-cancer treatment
Cumulative CIN2+ persistence | 24 months
  Proportion of participants with histologically confirmed CIN2+ up to 24 months after pre-cancer treatment
Cumulative CIN2+ persistence among participants with genotype-specific HPV persistence | 24 months
  Proportion of participants with histologically confirmed CIN2+ up to 24 months after pre-cancer treatment among participants with genotype-specific HPV persistence in first post-treatment cervical samples
Cumulative CIN2+ persistence among participants with HPV 16 or 18 | 24 months
  Proportion of participants with histologically confirmed CIN2+ up to 24 months after pre-cancer treatment among participants with HPV 16 or 18 in first post-treatment cervical samples
Cumulative CIN2+ persistence among participants with DNA hypermethylation | 24 months
  Proportion of participants with histologically confirmed CIN2+ up to 24 months after pre-cancer treatment among participants with DNA hypermethylation in first post-treatment cervical samples
Cumulative CIN2+ persistence among participants with any high-risk HPV | 24 months
  Proportion of participants with histologically confirmed CIN2+ up to 24 months after pre-cancer treatment among participants with any high-risk HPV in first post-treatment cervical samples
Association of baseline factors with CIN2+ persistence | 24 months
  Analysis of whether baseline factors-including CD4 cell count, HIV RNA viral load, HPV genotype, vaginal microbiome composition, sexually transmitted infections, cervical lesion grade, or type of pre-cancer treatment-are associated with cumulative CIN2+ persistence up to 24 months after pre-cancer treatment

SECONDARY OUTCOMES:
Association of baseline factors with genotype-specific HPV persistence | 24 months
  Analysis of whether baseline factors-including CD4 cell count, HIV RNA viral load, HPV genotype, vaginal microbiome composition, sexually transmitted infections, cervical lesion grade, or type of pre-cancer treatment-are associated with genotype-specific HPV persistence up to 24 months after pre-cancer treatment
Agreement beyond chance between HPV test results in paired cervical and urine samples | 0 months (baseline)
  Agreement between paired cervical and urine samples for HPV detection (type-specific and high-risk), measured before treatment and accounting for expected agreement by chance
Agreement beyond chance between HPV test results in paired cervical and urine samples | 6 months
  Agreement between paired cervical and urine samples for HPV detection (type-specific and high-risk), measured 6 months after treatment and accounting for expected agreement by chance
Agreement beyond chance between DNA methylation test results in paired cervical and urine samples | 0 months (baseline)
  Agreement between paired cervical and urine samples for DNA methylation testing, measured before treatment and accounting for expected agreement by chance
Agreement between beyond DNA methylation test results in paired cervical and urine samples | 6 months
  Agreement between paired cervical and urine samples for DNA methylation testing, measured 6 months after treatment and accounting for expected agreement by chance

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Pascoe, MD, Principal Investigator — Newlands Clinic Women's Health Centre
Locations (1):
- Women's Health Centre at Newlands Clinic, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No